#### Patient ID sticker

| INSERT RECRUITMENT SIT | Έ |
|------------------------|---|
| LOGO | |

# **PATIENT CONSENT FORM**

| STUDY: Prediction of venous thrombosis during chemotherapy-the PINPOINT study |
|---|
|---|

Recruitment Site: XXX. Site contact details to be inserted here

There are **two sections** in this form.

<u>Section 1</u> contains statements of understanding and asks you to tick each if you understand. Please ask any questions you may have when reading each of the statements.

<u>Section 2</u> asks for your consent to take part in this study. Please select either 'yes' or 'no' to indicate your choice.

<u>Section 3</u> asks for your consent sharing of the information and samples collected in this study with other researchers. Please select either 'yes' or 'no' to indicate your choice.

Thank you for participating. Please ask any questions if there is something you don't understand.

The end of this form is for the researchers to complete.

# If you wish to participate all boxes in section 1 must be ticked (V)

| 1. General Understanding | Tick |
|---|---|
| I confirm that I have read or had explained to me the Information Leaflet for<br>the above study. The information has been fully explained to me and I have<br>been able to ask questions, all of which have been answered to my<br>satisfaction. | |
| I understand that taking part in this study is entirely voluntary. I understand that not taking part will have no negative impact on me. | |
| I understand that I can leave this study at any time without giving a reason. I understand that leaving this study will not affect medical care, now or in the future. | |
| I understand that I will not be paid for taking part in this study or receive any benefits from taking part in this research study. | |
| I know how to contact the research team if I need to. | |
| By ticking each box above and choosing my options below <u>and</u> signing this docuparticipate in this study as described in the Participant Information Leaflet. | ıment I agree to |
| 2. Consent | |
| I agree to take part in this research study, having been fully informed of the risks and benefits in the participant information leaflet provided to me. | Yes No |



#### Patient ID sticker

INSERT RECRUITMENT SITE LOGO

| I agree to the use of blood samples and information about me (personal data) including information taken from my medical notes and records being used by the research team for this research study as described in the participant information leaflet. | Yes No |
|---|---|
| 3. Future Use of Samples and Data | Tick |
| I agree that information and samples collected for this study can be shared with other academic research institutions worldwide (research institutes, hospitals, not for profit organisations etc.) for research in the area of blood clotting and cancer research. All information and samples will only be shared subject to ethical approval and will comply with the GDPR. Any samples and information shared will use a unique code to protect your identity. | Yes No |
| I agree that information and samples- collected for this study can be shared with commercial companies carrying out health research worldwide for research in the area of blood clotting and cancer research. All information and samples will only be shared subject to ethical approval and will comply with the GDPR. Any information and samples shared will use a unique code to protect your identity. | Yes No |

I have ticked all the boxes which I agree to. By signing this document I agree to take part in this study as described in the patient information leaflet.

| Participant Name (Block Capitals) | Participant Signature | Date |
|---|---|---|
| Doctor/researcher name (Block Capitals) | Doctor/researcher Signature | Date |

### To be completed by the Principal Investigator or nominee.

I, the undersigned, have taken the time to fully explain to the above participant the nature and purpose of this study in a way that they could understand.

I have explained the risks and possible benefits involved. I have invited them to ask questions on any aspect of the study that concerned them.



# Patient ID sticker

INSERT RECRUITMENT SITE LOGO

I have given a copy of the participant information leaflet and consent form to the participant with contact details of the study team.

| Researcher name | | |
|--------------------------|--------|--------|
| Title and qualifications | | |
| Signature | | |
| Date | | |
| Date | | |
| Contact details | Email: | Phone: |

Copies to be created and retained: 1 for Participant, 1 for site/PI file and 1 for Hospital Records